CLINICAL TRIAL: NCT05238337
Title: A Phase 1, Open-label Study of the Absorption, Metabolism, and Excretion of [14C] PBI-200 Following a Single Oral Dose in Healthy Male Subjects
Brief Title: A Phase 1 Study of the Absorption, Metabolism, and Excretion of [14C] PBI-200
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pyramid Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBI-200-104
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Absorption, Metabolism and Excretion in Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-PBI-200 Treated (Experimental): [14C]-labeled PBI-200 will be administered as a single dose
  Interventions: Drug: [14C]-PBI-200

INTERVENTIONS:
Drug: [14C]-PBI-200 — [14C]-radio-labeled-PBI-200

SUMMARY:
This is a Phase 1, open-label non-randomized, single dose study in healthy male subjects.

DETAILED DESCRIPTION:
This is a Phase 1, open-label nonrandomized, single dose study in healthy male subjects to determine the absorption, metabolism, and excretion (AME) of [14C]-PBI-200

ELIGIBILITY:
Key Inclusion Criteria:

* Males, of any race, 18 to 65 years of age as of the dosing day.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive.
* Non-smoking/non-vaping, healthy, with no history of clinically relevant medical illness.

Key Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder.
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair will be allowed).

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Total Radioactivity in Urine and Feces | 28 days
Area Under the Concentration-Time Curve (AUC) of PBI-200 from time zero to infinity [AUC(0-inf)] | 28 days
Area Under the Concentration-Time Curve (AUC) of PBI-200 from time zero to the time of the last quantifiable concentration [AUC(0-tlast) | 28 days
Maximum Observed Concentration [C(max)] | 28 days
Time to Maximum Concentration [T(max)] | 28 days
Apparent Terminal Elimination Half-life [t(1/2)] | 28 days
Total Radioactivity in Plasma and Whole Blood | 28 days
Ratio for AUC(0-inf) Blood / Plasma | 28 days
Ratio for AUC(0-inf) Plasma PBI-200 / Total Radioactivity | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Pyramid Biosciences
Locations (1):
- Labcorp Clinical Research Unit Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No